CLINICAL TRIAL: NCT07287540
Title: Evaluation of the Effects of Anti-inflammatory Nutrition on the Outcomes of Non-surgical Periodontal Therapy in Individuals With Periodontitis
Brief Title: Anti-inflammatory Nutrition on the Outcomes of Non-surgical Periodontal Therapy
Status: Recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Hatice Yemenoğlu, Doctor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: Recep TayyipErdoğan University
Record Dates: First submitted 2025-11-17; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Periodontitis
Keywords: periodontitis; diet inflammatory index; anti-inflammatory nutrition
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Q3-1: Nonsurgical periodontal treatment and anti-inflammatory nutrition education
  Interventions: Other: non surgical periodontal trearment; Other: anti-inflammatory nutrition education
- Q3-2: Only nonsurgical periodontal treatment
  Interventions: Other: non surgical periodontal trearment
- Q4-1: Nonsurgical periodontal treatment and anti-inflammatory nutrition education
  Interventions: Other: non surgical periodontal trearment; Other: anti-inflammatory nutrition education
- Q4-2: Only nonsurgical periodontal treatment
  Interventions: Other: non surgical periodontal trearment

INTERVENTIONS:
Other: non surgical periodontal trearment — All participants will receive nonsurgical periodontal treatment
Other: anti-inflammatory nutrition education — Participants in Groups Q3-1 and Q4-1 will receive anti-inflammatory nutrition education
  Groups: Q3-1: Nonsurgical periodontal treatment and anti-inflammatory nutrition education; Q4-1: Nonsurgical periodontal treatment and anti-inflammatory nutrition education

SUMMARY:
This study aimed to determine the effect of anti-inflammatory nutrition on non-surgical periodontal treatment in individuals with periodontitis by evaluating gingival crevicular fluid (GCF) and serum biomarkers and clinical periodontal parameters.

A total of 100 volunteers identified as having a pro-inflammatory diet (Q3 and Q4) will be included in the study. Individuals will be assigned to two groups. These groups will then be further divided into two groups based on whether or not they will receive anti-inflammatory nutrition education. Group Q3-1 (n=25) will receive non-surgical periodontal treatment and anti-inflammatory nutrition education. Group Q3-2 (n=25) will receive only non-surgical periodontal treatment. Group Q4-1 (n=25) will receive non-surgical periodontal treatment and anti-inflammatory nutrition education. Group Q4-2 (n=25) will receive only non-surgical periodontal treatment. After the periodontal index measurements are completed, the patients will receive non-surgical periodontal treatment. GCF and serum samples, periodontal clinical parameters and Dietary Inflammatory Index will be collected 3 times: at baseline, 1.5 and 3 months after non-surgical periodontal treatment. Levels of interleukin (IL)-1β, IL-10, tumor necrosis factor (TNF)-α, total oxidant status (TOS), total antioxidant status (TAS), and C-reactive protein (CRP) will be assessed from these samples. This will investigate the role of anti-inflammatory nutrition in reducing periodontal inflammation and increasing treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy
* Not smoking
* Not using anti-inflammatory drugs in the last 3 months, antibiotics, or systemic corticosteroids in the last 6 months
* Not being pregnant or lactating
* Not having received periodontal treatment in the last 6 months
* Having at least 20 teeth in the mouth
* Being diagnosed with periodontitis by the investigator
* Having a dietary inflammatory index >0

Exclusion Criteria:

* Having a systemic disease
* Smoking
* Using anti-inflammatory drugs within the last 3 months, antibiotics within the last 6 months, or systemic corticosteroids
* Being pregnant or lactating
* Having received periodontal treatment within the last 6 months
* Having fewer than 20 teeth in the mouth
* No periodontitis

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study included individuals who applied to Recep Tayyip Erdogan University, Faculty of Dentistry, Department of Periodontology for treatment
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-02-21 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
periodontal pocket depth | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  It will be calculated by measuring the distance between the gingival margin and the pocket base. It will be measured from the six surfaces of each tooth and the average will be taken higher scores indicate worse outcome.
Clinical attachment loss | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  It will be calculated by measuring the distance between the cementoenemal border and the pocket base. It will be measured from the six surfaces of each tooth and the average will be taken higher scores indicate worse outcome.

SECONDARY OUTCOMES:
interleukin (IL)-1β level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  IL-1β levels will be measured with biochemical kits.
interleukin (IL)-10 level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  IL-10 levels will be measured with biochemical kits.
tumor necrosis factor (TNF)-α level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  TNF-α levels will be measured with biochemical kits.
serum total oxidant status (TOS) level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  TOS levels in serum will be measured with biochemical kits.
serum total antioxidant status (TAS) level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  TAS levels in serum will be measured with biochemical kits.
serum C-reactive protein (CRP) level | baseline, after nonsurgical periodontal treatment at 1.5 months, after nonsurgical periodontal treatment at 3 months.
  CRP levels in serum will be measured with biochemical kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No